CLINICAL TRIAL: NCT05747352
Title: Evaluation of the Glycemic Profile During the Ramadan Fasting in People With Type 1 Diabetes Treated With Closed-loop Hybrid Insulin System
Brief Title: Safety of Closed-loop Hybrid Insulin Administration During Ramadan Fasting in People Living With Type 1 Diabetes
Acronym: RAMDAM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0003
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Type1diabetes
Keywords: type1diabetes; the Ramadan fasting period; closed-loop hybrid insulin administration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: closed-loop hybrid insulin administration — observational non-interventional study

SUMMARY:
Fasting in Ramadan is not recommended for people with type 1 diabetes. The main risk associated with fasting is dysglycemia (hypoglycemia, hyperglycemia, diabetic ketosis) and dehydration. Nevertheless, whether or not to practice Ramadan remains a personal choice and many people living with diabetes choose to perform this fast with or without their physician's approval. The purpose of this prospective observational study is to evaluate the safety and efficacy of an closed-loop hybrid insulin system on glycemic parameters and the level of hypoglycemia in patients with type 1 diabetes who wished to fast during Ramadan.

DETAILED DESCRIPTION:
Primary objective: to evaluate the efficacy of an closed-loop hybrid insulin system on continuous glucose monitoring (CGM) glycemic parameters during the Ramadan fasting period Primary endpoint : to compare the time spent in the 3.9-10.0 mmol/l glucose target (TIR) from 30 days prior to the Ramadan fasting period to 30 days during the fasting period

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* type 1 diabetes for > 1 year
* on using closed-loop hybrid insulin administration
* scheduled Ramadan fasting
* patient put on using closed-loop hybrid insulin administration more than 2 months before the start of the Ramadan fast
* percentage of continuous glucose monitoring sensor wear > 70% in at least one of the two 30-day periods

Exclusion Criteria:

* patient put on using closed-loop hybrid insulin administration less than 2 months before the start of the Ramadan fast
* patient who is pregnant or wants to become pregnant immediately
* patient informed of the study who objected to the collection of his/her data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with type 1 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Glucose time | Day 30
  time spent in the 3.9-10.0 mmol/l glucose target (TIR)) in the Ramadan period

SECONDARY OUTCOMES:
Glucose time | Day 60
  The time spent in the 3.9-10.0 mmol/l glucose target (TIR)) in 30 days prior the Ramadan period
Glucose time | Day 30
  time spent below target 3.9 mmol/l
Glucose time | Day 60
  time spent below target 2.97 mmol/l, between 2.97 and 3.79 mmol/l, between 9.05 mmol/l and 12.5mmol/l and > 12.5 mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Dured DARDARI, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Outenah C, Ly Sall K, Penfornis A, Amadou C, Dardari D. Automated Insulin Delivery System: A Solution for Moderate to High-Risk Ramadan Fasting in People Living with Type 1 Diabetes. Diabetes Technol Ther. 2024 Nov;26(11):e881-e884. doi: 10.1089/dia.2024.0168. Epub 2024 Jul 17. PMID 38888435